CLINICAL TRIAL: NCT06740812
Title: Broadening Antiemetics Research by Comparing the Effectiveness of Fosaprepitant and Metoclopramide: A Randomized Control Trial
Brief Title: Broadening Antiemetics Research by Comparing the Effectiveness of Fosaprepitant and Metoclopramide
Acronym: BARF RCT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-16422
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Nausea and Vomiting; Nausea; Vomiting
Keywords: Signs and Symptoms, Digestive; Antiemetics; Autonomic Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Gastrointestinal Agents; Antipruritics; Dermatologic Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; Neurokinin-1 Receptor Antagonists; Fosaprepitant; Aprepitant; Dopamine Receptor Antagonist; Randomized Control Trial; Metoclopramide; Adults
MeSH Terms: conditions — Nausea; Vomiting; Signs and Symptoms, Digestive | interventions — fosaprepitant; Injections; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Intervention (Experimental): Fosaprepitant
  Interventions: Drug: Fosaprepitant for Injection
- Standard-of-Care Intervention (Active Comparator): Metoclopramide
  Interventions: Drug: Metoclopramide Injection

INTERVENTIONS:
Drug: Fosaprepitant for Injection — Fosaprepitant 150mg IV administered over 15 minutes
  Arms: Investigational Intervention
Drug: Metoclopramide Injection — Metoclopramide 10mg IV administered over 15 minutes
  Other Names: Reglan
  Arms: Standard-of-Care Intervention

SUMMARY:
The study team proposes a double-blind, comparative effectiveness, randomized controlled trial (RCT) to address the following goal: to determine the relative efficacy and adverse event profile of fosaprepitant compared to the standard of care antiemetic metoclopramide. Fosaprepitant and its active metabolite aprepitant are a relatively new class of antiemetic that exclusively acts in the central nervous system by blocking neurokinin (NK-1) which is a key signaling molecule in the centrally mediated aspects of the vomiting reflex. Currently, fosaprepitant and aprepitant both have only two United Stated Food and Drug Administration (USFDA) approved indications for nausea and vomiting: chemotherapy-induced and postoperative. Neurokinin inhibitors are highly effective and generally well-tolerated. Therefore, this class of medication may be a more appropriate medication for the millions of patients with nausea and vomiting that seek care in emergency departments (EDs). Intravenous fosaprepitant is converted to the active metabolite aprepitant on the order of minutes and is significantly cheaper to procure at this time.

DETAILED DESCRIPTION:
Nausea and vomiting (NV) are common and interrelated conditions. Approximately 50% of adults experience nausea in a given year while 30% of adults experience vomiting over the same period. Of this population of symptomatic individuals with NV, 25% of patients seek care in any healthcare delivery setting. Health Care Utilization Project (HCUP) data indicates that nearly 9.0 million patients seek care for NV in EDs each year in the United States.

Antiemetics are used to treat NV. Antiemetics currently utilized in the emergency department setting for NV do not always work on the first dose and have a plethora of side effects because of their peripheral mechanism of action outside of the vomiting reflex pathway in the central nervous system. These medications include ondansetron, promethazine, metoclopramide, olanzapine, haloperidol. Chief among these side effects is alteration of an aspect cardiac electrical signaling called the QT segment which represents the duration of ventricular contraction and relaxation. The QT segment is prolonged with commonly used antiemetics which can often be a prelude to cardiac dysrhythmias that are associated with mortality. As a result, patients with NV often have long length-of-stay (LOS) involving supportive care with intravenous fluids or empiric treatment with medications that can potentiate development of cardiac dysrhythmias. This is a problem in busy emergency departments (EDs) struggling to accelerate patient throughput in order to appropriately keep up with patient volume in an under-supplied hospital bed environment nationally.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old
* Present to ED for treatment of Nausea and/or vomiting as defined by the International Classification of Diseases (ICD-10) or identified by treating clinician

Exclusion Criteria:

* Pregnancy, desiring pregnancy, or lactating
* Antiemetic use or intravenous fluids prior to presenting to ED for evaluation and management
* Bradycardia (< 60 bpm heart rate)
* Prolonged QTc (greater than 490ms)
* Not conversant in English or Spanish
* Altered mental status
* Dementia
* Lack of phone for follow-up communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Sustained Nausea and Vomiting (NV) Relief | 2 hours (assessed at the 2-hour mark after administration of the intervention)
  The primary efficacy outcome for this study will be sustained relief from NV at 2 hours following medication administration. Sustained relief from NV will be determined by the intensity of nausea reported by patients following administration of antiemetic. Intensity of nausea will be reported as either "None", "Mild", "Moderate" or "Severe." The number/percentage of patients reporting each degree of nausea intensity at 2 hours will be summarized by study arm.
  Sustained relief of NV requires a patient to present with a nausea intensity of either "Severe" or "Moderate," which is then reduced by treatment to at least "Mild" or None," within 2 hours of medication administration without the use of any rescue medication. Patients who do not report an initial nausea intensity of either "Severe" or "Moderate" will not be assessed as they are not eligible for the study.
Development of New Symptom | 2 hours (assessed at the 2-hour mark after administration of the intervention)
  The primary tolerability outcome for this study will be the onset of any new symptoms within 2 hours after medication administration. Onset of symptoms will be assessed by asking patients if they developed any new symptoms after administration of the investigational medication. Symptoms will be elicited using an open-ended format. Patients who confirmed that they had experienced new symptoms will be asked to grade the severity of the new symptom(s) using the descriptors "Mild", "Moderate", or "Severe". The frequency and intensity of new symptoms will be summarized by study arm using basic descriptive statistics.

SECONDARY OUTCOMES:
Sustained NV Relief | 24 hours following medication administration
  Sustained relief from NV will be determined by the intensity of nausea reported by patients following administration of antiemetic. Intensity of nausea will be reported as either "None", "Mild", "Moderate" or "Severe." The number/percentage of patients reporting each degree of nausea intensity at 24 hours will be summarized by study arm.
  Sustained relief of NV requires a patient to present with a nausea intensity of either "Severe" or "Moderate," which is then reduced by treatment to at least "Mild" or "None," within 2 hours of medication administration AND maintained at "Mild" or "None" level for the entire 24-hour period following medication administration, without the use of rescue medication.
NV Relief | 24 hours (measured every 15 minutes for the first 2 hours, then hourly after that until final disposition; reassessed at 24 hours)
  Relief of NV over time will be determined by the intensity of nausea reported by patients following administration of antiemetic. Intensity of nausea will be reported as either "None", "Mild", "Moderate" or "Severe" and assessed every 15 minutes during the first 2 hours, then every hour after that up to 24 hours. The number/percentage of patients reporting each degree of nausea intensity at each timepoint will be summarized by study arm using basic descriptive statistics. Sustained relief of NV requires a patient to present with an initial nausea intensity of either "Severe" or "Moderate" and assessments will only be made in patients who did not need rescue medication.
NV Freedom | 24 hours (measured every 15 minutes for the first 2 hours, then hourly after that until final disposition; reassessed at 24 hours)
  Freedom from NV over time will be determined by the intensity of nausea reported by patients following administration of antiemetic. Intensity of nausea will initially be reported as either "None", "Mild", "Moderate" or "Severe" and assessed every 15 minutes during the first 2 hours, then every hour after that up to 24 hours. The number/percentage of patients reporting a nausea intensity of "None" will be summarized by study arm using basic descriptive statistics. Sustained freedom from NV requires a patient to present with an initial nausea intensity of either "Severe" or "Moderate" and assessments will only be made in patients who did not receive rescue medication.
Sustained NV Freedom | 24 hours following medication administration
  Sustained NV Freedom will be determined by the intensity of nausea reported by patients following administration of antiemetic. Intensity of nausea will initially be reported as either "None", "Mild", "Moderate" or "Severe." The number/percentage of patients reporting a nausea intensity of "None" will be summarized by study arm using basic descriptive statistics.
  Sustained NV Freedom requires a patient to present with a nausea intensity of either "Severe" or "Moderate," which is then reduced by treatment to "None" within 2 hours of medication administration AND maintained at the same ("None") level for the entire 24-hour period following medication administration, without the use of rescue medication.
Medication Preference | 24 hours
  Patient preference for receiving the same antiemetic medication as was administered during the study in the event of a subsequent episode of NV will be assessed during a follow-up phone call. Patients will be asked, "The next time you come to the ED for treatment of nausea and vomiting, do you want to receive the same medication again?" Patients will select from the following responses ("Yes," "No," or "Not sure"). Patient responses will be summarized and reported by study arm using basic descriptive statistics.
Duration of ED Stay | Initial presentation to disposition, approximately 4 hours
  Mean duration of ED stay, defined as the interval of time from initial presentation in ED to disposition, will be determined. ED durations will be summarized and reported by study arm using basic descriptive statistics. Prolonged LOS is generally associated with increased treatment complications and less favorable outcomes.

OTHER OUTCOMES:
Severity of Nausea | 24 hours (measured every 15 minutes for the first 2 hours, then hourly after that until disposition; reassessed at 24 hours)
  Severity of nausea will be evaluated based on responses to a visual analogue scale ranging from 0 to 100 (0 = no nausea, 100 = worst nausea possible). Mean scores will be summarized and reported by study arm. Higher scores are associated with increased severity of nausea.
QTc Interval (QT interval corrected for heart rate) | Prior to Intervention and at disposition, approximately 2 hours
  Mean QTc durations, as calculated from electrocardiogram (ECG) readings administered prior to receiving intervention, and at disposition, will be determined. Mean QTc durations will be summarized by study arm. Prolonged QT interval is commonly associated with antiemetics and can often be a prelude to cardiac dysrhythmias associated with mortality.
Need for rescue antiemetic medication | 2 hours (assessed at the 2-hour mark after administration of the intervention)
  The need for rescue antiemetic medication during the study will be assessed using a binary outcome (i.e., "Yes: or "No") to summarize whether additional dosing of antiemetic medication to treat nausea was needed. Results will be summarized by study arm using basic descriptive statistics.
Vomiting Episodes | Up to 24 hours
  The mean number of vomiting episodes per patient over the past 24 hours will be assessed and summarized by study arm.
Hospitalization | Up to 24 hours
  The percentage of patients who required hospitalization within 24 hours due to NV symptoms will be determined and summarized by study arm. Hospitalizations are associated with increased complications and less favorable outcomes.
Need for Fluid Treatment | 4 hours
  The percentage of patients treated with intravenous (IV) fluids will be determined and summarized by study arm. The need for IV fluids is associated with increased supportive care, increased hospital LOS and less favorable outcomes.
Mean Fluid Volume | 4 hours
  For patients requiring IV fluids, the mean per patient volume of IV fluids administered will be summarized and reported by study arm. The need for, and increased volumes of, IV fluids is associated with increased supportive care, increased hospital LOS and less favorable outcomes.
Revisit Rate to Emergency Department | 24 hours
  For purposes of this study, revisit rate will be defined as the number/percentage of participants requiring a revisit to the ED for additional evaluation and management of NV. Results will be summarized by study arm using basic descriptive statistics. More frequent revisit rates are associated with increased complications and less favorable outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mechanisms and Control of Emesis: A Satellite Symposium of the European Neuroscience Association: Proceedings of an International Meeting Held in Marseille (France), 4-7 September 1992. John Libbey Eurotext
- [Background] Singh P, Yoon SS, Kuo B. Nausea: a review of pathophysiology and therapeutics. Therap Adv Gastroenterol. 2016 Jan;9(1):98-112. doi: 10.1177/1756283X15618131. PMID 26770271
- [Background] Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Available from http://www.ncbi.nlm.nih.gov/books/NBK52651/ PMID 21413206
- [Background] Pourmand A, Mazer-Amirshahi M, Chistov S, Sabha Y, Vukomanovic D, Almulhim M. Emergency department approach to QTc prolongation. Am J Emerg Med. 2017 Dec;35(12):1928-1933. doi: 10.1016/j.ajem.2017.08.044. Epub 2017 Aug 24. PMID 28855066
- [Background] Franklin BJ, Vakili S, Huckman RS, Hosein S, Falk N, Cheng K, Murray M, Harris S, Morris CA, Goralnick E. The Inpatient Discharge Lounge as a Potential Mechanism to Mitigate Emergency Department Boarding and Crowding. Ann Emerg Med. 2020 Jun;75(6):704-714. doi: 10.1016/j.annemergmed.2019.12.002. Epub 2020 Jan 23. PMID 31983501
- [Background] Aapro M, Carides A, Rapoport BL, Schmoll HJ, Zhang L, Warr D. Aprepitant and fosaprepitant: a 10-year review of efficacy and safety. Oncologist. 2015 Apr;20(4):450-8. doi: 10.1634/theoncologist.2014-0229. Epub 2015 Mar 20. PMID 25795636
- [Background] Langford P, Chrisp P. Fosaprepitant and aprepitant: an update of the evidence for their place in the prevention of chemotherapy-induced nausea and vomiting. Core Evid. 2010 Oct 21;5:77-90. doi: 10.2147/ce.s6012. PMID 21042544
- [Background] Furyk JS, Meek RA, Egerton-Warburton D. Drugs for the treatment of nausea and vomiting in adults in the emergency department setting. Cochrane Database Syst Rev. 2015 Sep 28;2015(9):CD010106. doi: 10.1002/14651858.CD010106.pub2. PMID 26411330
- [Background] Yang Y, Yang N, Wu L, Ouyang Q, Fang J, Li J, Liao W, Cai K, Huang J, Li J, Zhang Y, Wang X, Zhang H, Xu N, Zhao Q, Hu X, Li W, Zhong W, Zhong D, Cheng G, Ye S, Zhong M, Wang D, Liu H, Zheng J, Liu X, Xu H, Zhang L. Safety and efficacy of aprepitant as mono and combination therapy for the prevention of emetogenic chemotherapy-induced nausea and vomiting: post-marketing surveillance in China. Chin Clin Oncol. 2020 Oct;9(5):68. doi: 10.21037/cco-20-160. PMID 33161724
- [Background] Braude D, Soliz T, Crandall C, Hendey G, Andrews J, Weichenthal L. Antiemetics in the ED: a randomized controlled trial comparing 3 common agents. Am J Emerg Med. 2006 Mar;24(2):177-82. doi: 10.1016/j.ajem.2005.08.017. PMID 16490647
- [Background] Cham S, Basire M, Kelly AM. Intermediate dose metoclopramide is not more effective than standard dose metoclopramide for patients who present to the emergency department with nausea and vomiting: a pilot study. Emerg Med Australas. 2004 Jun;16(3):208-11. doi: 10.1111/j.1742-6723.2004.00588.x. PMID 15228463